CLINICAL TRIAL: NCT06467448
Title: Comparing Train-of-Four Recovery in the Adductor Pollicis Versus the Adductor Digiti Minimi in Elective Surgery Patients Using EMG
Brief Title: Comparing Train-of-Four Recovery in the Adductor Pollicis Versus the Adductor Digiti Minimi in Elective Surgery Patients
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 24-1013
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Adductor Pollicis EMG: The Train of Four Ratio will be recorded at 90% as a time and as a reference point
  Interventions: Device: EMG Assessement of Recovery of Neuromuscular Function
- Adductor Digiti Minimi: The Train of Four Ratio will be recorded when the adductor pollicis ratio reads 90%
  Interventions: Device: EMG Assessement of Recovery of Neuromuscular Function

INTERVENTIONS:
Device: EMG Assessement of Recovery of Neuromuscular Function — EMG Train of Four Assessment of Recovery of Neuromuscular Function

SUMMARY:
The train-of-four (TOF) ratio is a quantitative measure used in anesthesia to assess the degree of neuromuscular blockade induced by neuromuscular blocking agents during surgical procedures. Current American Society of Anesthesiologists guidelines recommend monitoring the TOF ratio to guide the administration and reversal of NMBAs, with a target ratio of 0.9 or higher at adductor pollicis muscle indicating adequate reversal and restoration of neuromuscular function.

This proposed study aims to observe and compare the TOF ratio between two different muscles of the hand: adductor pollicis and adductor digiti minim using anesthesia monitors on both of their arms during recovery of neuromuscular function. Surgery and anesthesia will occur per standard of care.

DETAILED DESCRIPTION:
The study population will enroll adult patients (>18) who will receive non-depolarizing neuromuscular blocking drugs as part of a routine general anesthetic and who will have monitoring of their recovery from neuromuscular block performed using the Tetragraph (Senzime Sweden). Patients with upper limb weakness, neurological deficits, and inability to use the other arm to record the second EMG recording will be excluded.

Procedures (methods):

Adult patients undergoing general anesthesia with the use of muscle relaxants will have anesthesia monitors on both of their arms. On one arm, the study sticky pad will be placed on the forearm and over the base of the little finger. On the other arm, the standard monitor is placed on the forearm and over the base of the thumb.

To identify pre-operative patients, an EPIC report will be utilized to screen for eligible participants. Patients will be contacted via phone by a research team member the day before their procedure and enrolled. Informed consent will be formally obtained on the day of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Surgery and general anesthesia with administration of non depolarizing neuromuscular blocking drug

Exclusion Criteria:

* neuromuscular disease or weakness of one of upper limbs.
* Inability to use one of subjects arms to record neuromuscular monitor.
* Contraindication to administration or allergy to non depolarizing neuromuscular blocking drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consented patients undergoing general anesthesia with an endotracheal tube and non depolarizing muscle relaxants and objective monitoring of train of four.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in Measured Recovery of Train of Four at Adductor Pollicis and Adductor Digiti Minimi | All assessments are intraoperative and complete in one day
  The train of four ratio at the digiti minimi will be recorded when the adductor pollicis ratio reads 90 percent

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Grant, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No